CLINICAL TRIAL: NCT01164293
Title: Prevalence of Positive Reactions in Atopy Patch Test in Children With Food Allergy-related Gastrointestinal Symptoms
Brief Title: Atopy Patch Test in Children With Food Allergy-related Gastrointestinal Symptoms
Acronym: APT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 079/2553(EC1)
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Food Allergy
Keywords: Atopy patch test
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atopy patch test (Experimental): Atopy patches were applied on food allergy patient's back for 48 hrs then the patches were removed. Reaction was evaluated at 48 and 72 hrs after applying atopy patch test
  Interventions: Device: Atopy patch test with food allergen

INTERVENTIONS:
Device: Atopy patch test with food allergen — Atopy patches used with food lyophilized allergen and commercial allergen were placed on back of subjects for 48 hrs then atopy patches were taken off. Subjects should return to evaluate the reaction one day later (72 hr after applying atopy patch test)
  Other Names: Fin chamber

SUMMARY:
Positive reactions in Atopy patch test in children with food allergy-related gastrointestinal symptoms

DETAILED DESCRIPTION:
The prevalence of food allergy seems to be increasing, which might explain the increased demand for reliable evaluation of patients with suspected food-related gastrointestinal symptoms. Little is known about the diagnostic accuracy of atopy patch tests(APT) in the clinical practice. APT seems to have a better specificity than the IgE methods and seems to reflect late-phase clinical reactions.The aims of this study were to evaluate:

(i) The prevalence of positive reaction of APTs for food allergy-related gastrointestinal diseases. (ii)Positive reaction of APT compare with skin prick test. (iii)Positive reaction of APT using lyophilized food vs commercially available food extracts. (iv)Side effect or adverse events of APT

ELIGIBILITY:
Inclusion Criteria:

* Patients who had history of suspected food allergy-related gastrointestinal symptoms eg. nausea and vomiting, diarrhea, abdominal pain or hematochezia after ingesting some food.
* Age 1 month-18 yrs
* Elimination diet was done at least 7 days before starting the study
* Written informed consent was obtained from the parents of each child enrolled in the study

Exclusion Criteria:

* Who have dermographism
* Who have chronic disease eg. autoimmune disease, immune deficiency, cancer or allergic disease
* Pregnant women
* Who have severe eczema
* Who receive antihistamine, topical steroid and systemic steroid > 20 mg/day withiin 7 days prior study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of positive reaction in APT in children with food allergy-related gastrointestinal symptoms | 3 days
  To evaluate (i) The prevalence of positive reaction of APTs for food allergy-related gastrointestinal diseases. (ii)Positive reaction of APT compare with skin prick test.

SECONDARY OUTCOMES:
Comparisons atopy patch test reaction between lyophilized allergen and commercial allergen | 3 days
  To evaluate (iii)Positive reaction of APT using lyophilized food vs commercially available food extracts. (iv)Side effect or adverse events of APT

CONTACTS AND LOCATIONS:
Overall Officials: Nualanong Visitsunthorn, MD, Study Director — Mahidol University
Locations (1):
- Department of Pediatrics, Siriraj hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Visitsunthorn N, Chatpornvorarux S, Pacharn P, Jirapongsananuruk O. Atopy patch test in children with atopic dermatitis. Ann Allergy Asthma Immunol. 2016 Dec;117(6):668-673. doi: 10.1016/j.anai.2016.09.446. PMID 27979025